CLINICAL TRIAL: NCT00873704
Title: Supplemental Postoperative Oxygen and the Risk of Surgical Wound Infection in a Vascular Surgery Population: A Randomized Controlled Trial
Brief Title: Supplemental Oxygen in Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKCH-Surg-003
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Surgical Wound Infection; Vascular Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): recieves supplemental oxygen postoperatively
  Interventions: Other: supplemental postoperative oxygen
- 2 (No Intervention): treated as usual without supplemental oxygen

INTERVENTIONS:
Other: supplemental postoperative oxygen
  Arms: 1

SUMMARY:
The purpose of this study was to test the hypothesis that supplemental postoperative oxygen reduces the risk of surgical wound infection in patients following lower limb vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* lower limb vascular surgery

Exclusion Criteria:

* COPD
* sPO2 less than 90%

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
surgical wound infection | 30 days

CONTACTS AND LOCATIONS:
Locations (6):
- Finland (6):
  - North Karelia Central Hospital, Joensuu
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - South Karelia Central Hospital, Lappeenranta
  - Central Hospital of Mikkeli, Mikkeli
  - Lapland Central Hospital, Rovaniemi

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Turtiainen J, Saimanen EI, Partio TJ, Makinen KT, Reinikainen MT, Virkkunen JJ, Vuorio KS, Hakala T. Supplemental postoperative oxygen in the prevention of surgical wound infection after lower limb vascular surgery: a randomized controlled trial. World J Surg. 2011 Jun;35(6):1387-95. doi: 10.1007/s00268-011-1090-y. PMID 21476113